CLINICAL TRIAL: NCT06074575
Title: The Effect of Positive and Negative Emotions on Mechanical Pain Thresholds: a Randomized Controlled Trial
Brief Title: Do Emotions Affect Mechanical Pain Thresholds?
Acronym: DEAMPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linnaeus University (Other)
Responsible Party: Principal Investigator, Helena Gunnarsson, Principal Investigator, Linnaeus University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-03968-01
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2023-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Within-subjects design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Negative emotional condition (Experimental): The participant will watch a short video-clip with negative emotional content.
  Interventions: Behavioral: Emotion induction
- Positive emotional condition. (Experimental): The participant will watch a short video-clip with positive emotional content.
  Interventions: Behavioral: Emotion induction
- Neutral condition. (Experimental): The participant will watch a short video-clip with neutral emotional content.
  Interventions: Behavioral: Emotion induction
- Control condition. (Experimental): The participant will not watch a video-clip, but will wait without specific instructions about what to think about.
  Interventions: Behavioral: Emotion induction

INTERVENTIONS:
Behavioral: Emotion induction — The participants will receive different emotion inductions through short video clips.

SUMMARY:
The purpose of this study is to investigate if different emotional states could influence mechanical pain thresholds.

DETAILED DESCRIPTION:
Participants will be randomized into 4 different groups watching different short video-clips (2.20 min). The negative emotions group will watch an uncomfortable short video containing violence and blood, the positive emotions group will watch a video containing a stand-up comedy show, the neutral emotions group will watch a video with Swedish nature, and the control group will just wait for 2.20 min, without any instructions about what to think about. Pressure pain thresholds will be measured with an algometer before and after the video-clip interventions.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years of age, fluent in Swedish.

Exclusion Criteria:

* Pain anywhere in body during the test session, known neurological disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold | Measurements will be conducted at the test session, which will have a duration of approximately 20 minutes for each participant.
  Pressure pain threshold value after each different emotion intervention and control compared to before each emotion intervention and control.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Gunnarsson, PhD, Principal Investigator — Linnéuniversitetet
Locations (1):
- Helena Gunnarsson, Vaxjo, Kronoberg County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Data is available after study completion.
Supporting Information: SAP
Time Frame: The data will be available after study completion.
Access Criteria: The data is anonymous and is therefore freely available.